CLINICAL TRIAL: NCT05355844
Title: Can Benzoyl Peroxide Decrease the Burden of Cutibacterium Acnes in Primary Spine and Shoulder Surgery? Prospective Randomized Study
Brief Title: Cutibacterium Acnes in Deep Tissues in Primary Spine and Shoulder Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital del Mar (Other)
Responsible Party: Principal Investigator, Carlos Torrens, Clinical Professor, Hospital del Mar
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2022/10272
Record Dates: First submitted 2022-04-26; First posted 2022-05-02 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Rotator Cuff Tear Arthropathy; Spine Degeneration
MeSH Terms: conditions — Rotator Cuff Tear Arthropathy | interventions — Benzoyl Peroxide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients without Benzoyl peroxide (Sham Comparator)
  Interventions: Drug: Benzoyl peroxide
- Patients with Benzoyl peroxide (Experimental)
  Interventions: Drug: Benzoyl peroxide

INTERVENTIONS:
Drug: Benzoyl peroxide — Benzoyl peroxide application in the incision area before surgery

SUMMARY:
Obtain deep tissue samples from patients undergoing primary prosthetic surgery of the shoulder and patients undergoing primary instrumented surgery of the spine. Patients will be randomized to receive benzoyl peroxide 3 days prior to surgery.

DETAILED DESCRIPTION:
Shoulder prosthetic surgery as well as interventional surgery on the spine are commonly contaminated by Cutibacterium Acnes. Although the significance of this contamination is unknown, it represents a cause for concern since in some patients, contaminating Cutibacterium Acnes from surgery may develop long-term infection of the implant. Unlike knee and hip surgeries, where the most common infection-causing germs are Staphylococcus aureus, in shoulder and spine surgery, Cutibacterium Acnes represents one of the germs most frequently associated with infections. peri implant. Skin preparation with chlorhexidine as well as antibiotic prophylaxis with cefazolin have been shown to be ineffective in eradicating Cutibacterium Acnes. Recently, different studies support the use of benzoyl peroxide in topical application, to reduce the load of Cutibacterium acnes on the skin. Despite this, it has not been shown to reduce the rate of infection, nor to reduce the phylotypes of Cutibacterium acnes associated with peri-implant infections (IA, IB and II).

Obtain deep tissue samples from patients undergoing primary prosthetic surgery of the shoulder and patients undergoing primary instrumented surgery of the spine. Patients will be randomized to receive benzoyl peroxide 3 days prior to surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients > 18 yrs.
* Primary prosthetic shoulder surgery.
* Instrumented primary surgery of the spine.

Exclusion Criteria:

* active infection.
* previous surgeries.
* interventionism prior to surgery in the last 6 months (infiltrations, arthro-CT, arthro-MRI)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2023-05 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Cutibacterium acnes | 2 weeks
  isolation of Cutibacterium acnes in the deep tissues

IPD SHARING:
Plan to Share IPD: No